CLINICAL TRIAL: NCT05071066
Title: Evaluation for the Pilot Scheme on New Service Protocol for Attention Deficit/Hyperactivity Disorder With Comorbidity ("ADHD+"): A Randomized Waitlist-controlled Trial
Brief Title: New Service Protocol for Attention Deficit/Hyperactivity Disorder With Comorbidity: A Randomized Waitlist-controlled
Acronym: ADHD+
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Yi-Nam Suen, Research Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ADHD+HK
Record Dates: First submitted 2021-09-27; First posted 2021-10-07 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-09

CONDITIONS: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group-based ADHD+ Treatment (Experimental): This randomized controlled trial (RCT) will run in multi-sites including 5 non-governmental organizations (NGOs) in Hong Kong. Core treatment components are developed by an expert group comprised of psychiatrists and clinical psychologists including internet use/addiction intervention, cognitive training, etc.
  The main intervention lasts for 3 months, and the booster intervention lasts for another 3 months.
  Interventions: Other: ADHD+
- wait-list control group (Other): For participants in the waiting list control group, they will receive 1-3 hours psychoeducation during the 3 months wait period. Appropriate intervention will be offered after the treatment group.
  Interventions: Other: ADHD+

INTERVENTIONS:
Other: ADHD+ — The group-based intervention is designed to reduce participants' ADHD and related symptoms. The content of the treatment will follow an established manual which is developed by an expert group comprised of psychiatrists and clinical psychologists. Core treatment components include internet use/addiction intervention, cognitive training, emotion management, social skills training, occupational training, emotion support/befriending, parenting training, and career guidance.
  The main intervention lasts for 3 months, and the booster intervention lasts for another 3 months. The post- intervention assessments (3-month [T1], and 6-month [T2]) will be administered to all participants. During the period of intervention, all participants shall be clean from other forms of interventions to reduce any other possible confounders.

SUMMARY:
The proposed study is to be carried out in 2021 - 2024 with youths aged 6 - 15 in Hong Kong. This is a randomized waitlist-controlled trial that aims to examine the effectiveness of the ADHD+ new service protocol. This ADHD+ new service protocol intervention will be delivered for 6 months in the format of groups by frontline social workers trained by professional clinicians including clinical psychologists and psychiatrists. It is designed to reduce ADHD and related symptoms in individuals aged between 6 and 15 years.

Core treatment components include internet use/addiction intervention, cognitive training, emotion management, social skills training, occupational training, emotion support/befriending, parenting training, and career guidance. It is hypothesized that youths receiving the intervention will have reduced ADHD and related symptoms when compared with controls.

Findings will allow the investigators to better understand the effectiveness of the new ADHD+ service; and in the long run, the service model can be generalized to community based early interventions for other uncomplicated mental disorders.

ELIGIBILITY:
Inclusion Criteria:

* children, adolescent and young adults (Aged 6-15);
* have sufficient proficiency in Chinese to understand verbal instructions and give informed consent;
* clinically significant mild to moderate ADHD syndromes requiring intervention;
* without learning disabilities and intelligence quotient (IQ) score not lower than 70;
* are "more likely to commit time in the projects" for reasons such as intention to treat and
* receiving the New ADHD+ service.

Exclusion Criteria:

* known diagnosis of intellectual disability;
* not reaching syndrome diagnostic threshold for ADHD;
* already receiving medical interventions / treatments at Hospital Authority (HA) and/or private sector;
* known psychiatric diagnosis (stabilized diagnosis and treatment);
* current or active suicidal ideation or attempts;
* have received structured psychosocial intervention for more than 3 contact hours (for waitlist group); and
* refusal to give consent.

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2021-12-20 (Actual); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
The change of overall ADHD and related symptoms | From Time 0 (Baseline) to Time 1 (post-intervention 3-month) to Time 2 (post-intervention 6-month)
  Measured by Strengths and Weaknesses of ADHD-symptoms and Normal-behaviors questionnaire (SWAN) (for service users under 18 years old) (parent report). The scale has 18 items, each rated from -3 to 3 following 7-point Likert scale. Higher scores indicate greater symptomology
The change of difficult behavior in service users | From Time 0 (Baseline) to Time 1 (post-intervention 3-month) to Time 2 (post-intervention 6-month)
  Measured by Strengths and Difficulties Questionnaires (SDQ) [children version]. The scale has 25 items, each rated from 0 - 2. Higher score indicate more difficult behaviors.

CONTACTS AND LOCATIONS:
Overall Officials: YI Nam Suen, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No